CLINICAL TRIAL: NCT02285608
Title: Partnership in Medication Management (PIMM): The Effects of One-on-one Medication Training on Medication Adherence in Patients With Mood Disorders
Brief Title: Partnership in Medication Management (PIMM) in Patients With Mood Disorders
Acronym: PIMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PIMM MDP; PIMM Mood Disorders Program (Other Grant/Funding Number: Mood Disorders Program, St. Joseph/s Healthcare Hamilton)
Record Dates: First submitted 2014-10-28; First posted 2014-11-07 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Medication adherence; Patient education; Mood disorders; Economic assessment; Mixed methods
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Medication Adherence; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PIMM/SAM (Experimental): Partnership in Medication Management (PIMM): The nurse and the attending physician will meet with the patient and ask how s/he administers medication at home (i.e., blister pack). Initial education session: the nurse will teach the patient about his/her medications, dosage, purpose, when and how to take them. Nurse and patient will establish reminders to take his/her medication. Following the education session, patients will be required to notify the nurse when it is time to take their medications, where their medications are, dosage, purpose and side effects. Self-Administered Medication (SAM): Patients will transition to SAM once the clinical team feels that no further medication changes are required. SAM is also the model that the participants will follow after discharge.
  Interventions: Other: PIMM/SAM
- Standard Prescribing Practice(SPP) (No Intervention): Standard prescribing practice (SPP): medication administration will proceed as standard practice. Patients will not receive a personalized medication training. The nurse will administer the patient's medications. However, patients are encouraged to ask any questions regarding his/her medications.Patients will not be provided with any tool to help them to remember when to take their medications. The nurse will record the patient's knowledge regarding his/her medications.

INTERVENTIONS:
Other: PIMM/SAM — The PIMM program will include education to improve patients' knowledge regarding their medication's purpose, dosage, benefits, and side effects. The program will also include tools like a checklist or alarm clock to remind patients of when and how to take their medication. Furthermore, the program will contain an interactive listening period where healthcare professionals involved in medication dispensing will listen to patients' concerns, questions and thoughts regarding their medications.
  Other Names: Partnership in Medication Management
  Arms: PIMM/SAM

SUMMARY:
Investigators are doing this study to examine if a new personalized education program for patients with mood disorders (depression and bipolar disorders) will help them take their medications as prescribed by doctors. Investigators will teach patients about how, when and why it is important for them to take their medications as prescribed. Also, investigators will ask patients why they do not take medications as prescribed. Furthermore, investigators will examine whether our education program might save money if it prevents problems related to not taking medication.

DETAILED DESCRIPTION:
The efficacy of anti-depressants or lithium reported in clinical trials differs from clinical experience. Various factors such as non-adherence to treatment and poor tolerability to medications have been related to treatment non-response or treatment failure in mood disorders (major depressive disorder and bipolar disorder). Premature discontinuation of treatment for mood disorders is common. The long treatments, the patients' beliefs about medications, the lack of knowledge about the medication/treatment purpose, benefits, dosage, and side effects and the relationship between patient and healthcare providers affect treatment continuation.

Investigators are proposing a sequential explanatory mixed methods study to investigate a novel program for medication training in persons with mood disorders. The ultimate purpose of the program is to improve medication adherence in these persons. The primary component of the present study will be quantitative, i.e., a randomized controlled trial with 12 months of follow-up to examine the effect of one-on-one medication training, including the use of a checklist system, on medication adherence in patients with mood disorders. The training program will include education to improve patients' knowledge regarding their medication's purpose, dosage, benefits, and side effects. The program will also include tools like a checklist or alarm clock to remind patients of when and how to take their medication. Furthermore, the program will contain an interactive listening period where healthcare professionals involved in medication dispensing will listen to patients' concerns, questions and thoughts regarding their medications. To the best of the investigators' knowledge, no research has comprehensively examined whether one-on-one medication training, as described above, may improve medication adherence in patients with mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the inpatient clinic of the Mood Disorders Program, St. Joseph's Healthcare Hamilton
* with a primary diagnosis of bipolar disorder I or II, or major depressive disorder
* able to speak, read, and understand English.

Exclusion Criteria:

* cut off score on Montreal Cognitive Assessment (MOCA; clinical judgement)
* significant suicidal or homicidal risk
* a medical condition/treatment known to affect the brain
* acquired brain injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-11 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Medication adherence measured by the Medication Adherence Rating Scale (MARS). | Change from baseline in the Medication Adherence Rating Scale at 2 days before discharge and 1 week, 1 month, 3 months, 6 months and 12 months post-discharge
  Medication adherence measured by the Medication Adherence Rating Scale (MARS). We will measure medication adherence at baseline and each follow up

SECONDARY OUTCOMES:
Time to re-hospitalization | First time re-hospitalization any point during the 12-month follow-up period
  Investigators will compare the time to re-hospitalization between each study group.
Costs of re-hospitalization | First time re-hospitalization any point during the 12-month follow-up period
  Investigators will adopt a healthcare system perspective and compare the costs of first re-hospitalization between each study group. When a participant is re-hospitalized for the first time at any point during the 12-month follow-up period, investigators will conduct a chart review of the entire re-hospitalization to identify all of the direct and indirect medical resources consumed during this re-hospitalization. The chart review will cover the entire length of the re-hospitalization, even if this length exceeds the 12-month follow-up period for the participant in question.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Oremus, MD, PhD(c), Principal Investigator — McMaster University; Sharon Simmons, RN,BScN,CPMHNc, Principal Investigator — St. Joseph's Healthcare Hamilton; Margaret C McKinnon, PhD,C.Psych., Principal Investigator — McMaster University
Locations (1):
- Mood Disorders Program, St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] The World Health Organization.The global burden of disease: 2004 update, Table A2: Burden of disease in DALYs by cause, sex and income group in WHO regions, estimates for 2004. Geneva, Switzerland, 2008 (accessed on: March 6, 2014).
- [Background] Health Canada. A Report on Mental Illnesses in Canada. Ottawa: Health Canada, 2002.
- [Background] World Health Organization. Adherence to Long- Term Therapies: Evidence for Action. Geneva, Switzerland: World Health Organization, 2003.
- [Background] Rosa AR, Marco M, Fachel JM, Kapczinski F, Stein AT, Barros HM. Correlation between drug treatment adherence and lithium treatment attitudes and knowledge by bipolar patients. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jan 30;31(1):217-24. doi: 10.1016/j.pnpbp.2006.08.007. Epub 2006 Sep 18. PMID 16982121
- [Background] Nemeroff CB, Heim CM, Thase ME, Klein DN, Rush AJ, Schatzberg AF, Ninan PT, McCullough JP Jr, Weiss PM, Dunner DL, Rothbaum BO, Kornstein S, Keitner G, Keller MB. Differential responses to psychotherapy versus pharmacotherapy in patients with chronic forms of major depression and childhood trauma. Proc Natl Acad Sci U S A. 2003 Nov 25;100(24):14293-6. doi: 10.1073/pnas.2336126100. Epub 2003 Nov 13. PMID 14615578